CLINICAL TRIAL: NCT00857402
Title: Arginine Rich Food Supplementation as an Adjuvant Treatment Against Tuberculosis
Brief Title: Arginine as an Adjuvant Treatment Against Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University of Gondar (Other); Kalmar County Hospital (Other)
Responsible Party: Thomas Schön, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ArgII; HLF_20060246
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Tuberculosis; HIV
Keywords: Arginine; Nitric oxide; Peanuts; Sedimentation rate
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peanuts (Active Comparator)
  Interventions: Dietary Supplement: Peanuts
- Daboqolo (Active Comparator)
  Interventions: Dietary Supplement: Daboqolo

INTERVENTIONS:
Dietary Supplement: Peanuts — 30g of peanuts daily for 4 weeks (directly observed). This dose of peanuts is equivalent to 1 gram of arginine.
  Arms: Peanuts
Dietary Supplement: Daboqolo — 30g of Daboqolo per os daily for 4 weeks (given supervised). 30g of Daboqolo is equivalent to 0.1 g of arginine.
  Arms: Daboqolo

SUMMARY:
The purpose of this study was to investigate if adjuvant treatment with arginine (the substrate for nitric oxide production) rich food supplements could improve clinical outcome in patients with smear positive tuberculosis by affecting nitric oxide production.

DETAILED DESCRIPTION:
Tuberculosis (TB) is disease of increased global public health importance. Because of emerging multi drug resistance and the long treatment duration there is a need to optimize the current chemotherapy. Host immunity is important in determining the susceptibility and outcome of disease as could be exemplified by co infection with HIV which dramatically increases the risk to develop TB.

Previous results from our group and others show that nitric oxide produced by activated macrophages from arginine might be important to control the disease. However, the relative importance of nitric oxide in human TB has been debated. In a previous study in Gondar, Ethiopia, we observed an effect of adjuvant treatment with arginine capsules on sputum smear conversion and reduction of cough. In this study we wanted to test the hypothesis based on previous observations that an arginine rich food supplementation might enhance clinical improvement in patients with smear positive tuberculosis and if this effect could be due to increased nitric oxide production.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent to take part in the study
* Previously untreated and newly diagnosed smear positive Tb patients according to the WHO definitions

Exclusion Criteria:

* Hospitalization
* Pregnancy
* Known allergy against peanuts
* Chronic or acute disease other than tuberculosis/HIV

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Final outcome according to WHO | 8 months

SECONDARY OUTCOMES:
Change in Chest X-ray pattern from baseline to 2 months | 2 months
Levels of exhaled and urinary nitric oxide | First week, week 2, week 8, and month 5
Weight gain from baseline until 2 months | 2 months
Sedimentation rate | 2 months
Sputum smear conversion | 2 months
Reduction of cough from baseline to 2 months | 1 and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schön, MD PhD, Principal Investigator — Linkoeping University; Sven Britton, Professor, Study Director — Karolinska Institutet; Tommy Sundqvist, Professor, Study Chair — Linkoeping University, Sweden
Locations (1):
- Gondar University, DOTS-center, Gondar, Region 3, Ethiopia, Gondar, Ethiopia

REFERENCES:
- [Background] Schon T, Wolday D, Elias D, Melese E, Moges F, Tessema T, Stendahl O, Sundqvist T, Britton S. Kinetics of sedimentation rate, viral load and TNF-alpha in relation to HIV co-infection in tuberculosis. Trans R Soc Trop Med Hyg. 2006 May;100(5):483-8. doi: 10.1016/j.trstmh.2005.07.018. Epub 2005 Oct 20. PMID 16242741
- [Background] Schon T, Elias D, Moges F, Melese E, Tessema T, Stendahl O, Britton S, Sundqvist T. Arginine as an adjuvant to chemotherapy improves clinical outcome in active tuberculosis. Eur Respir J. 2003 Mar;21(3):483-8. doi: 10.1183/09031936.03.00090702. PMID 12662006
- [Background] Wang CH, Liu CY, Lin HC, Yu CT, Chung KF, Kuo HP. Increased exhaled nitric oxide in active pulmonary tuberculosis due to inducible NO synthase upregulation in alveolar macrophages. Eur Respir J. 1998 Apr;11(4):809-15. doi: 10.1183/09031936.98.11040809. PMID 9623681
- [Result] Idh J, Westman A, Elias D, Moges F, Getachew A, Gelaw A, Sundqvist T, Forslund T, Alemu A, Ayele B, Diro E, Melese E, Wondmikun Y, Britton S, Stendahl O, Schon T. Nitric oxide production in the exhaled air of patients with pulmonary tuberculosis in relation to HIV co-infection. BMC Infect Dis. 2008 Oct 24;8:146. doi: 10.1186/1471-2334-8-146. PMID 18950489
- [Derived] Schon T, Idh J, Westman A, Elias D, Abate E, Diro E, Moges F, Kassu A, Ayele B, Forslund T, Getachew A, Britton S, Stendahl O, Sundqvist T. Effects of a food supplement rich in arginine in patients with smear positive pulmonary tuberculosis--a randomised trial. Tuberculosis (Edinb). 2011 Sep;91(5):370-7. doi: 10.1016/j.tube.2011.06.002. Epub 2011 Aug 2. PMID 21813328